CLINICAL TRIAL: NCT00735956
Title: PARTNER: The Underage Drinking: Building Health Care System Research
Brief Title: PARTNER Recruitment and Brief Intervention Pilot Study
Acronym: PARTNER
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Robert L Hubbard, Ph.D., Duke University / NDRI
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00006998
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Last update posted 2010-08-23 (Estimated); Status verified 2010-08

CONDITIONS: Alcohol Abuse
Keywords: Screening; Brief Intervention
MeSH Terms: conditions — Alcoholism | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Counseling — Handouts, referrals and brief counseling sessions are given after determination of early alcohol abuse has been assessed.
  Other Names: CRAFFT; Other Shared Items Proposal

SUMMARY:
Purpose of the study:

This is a pilot randomized controlled trial to identify methods of involving underage youth in interventions to reduce alcohol use through the primary health care system. The trial will compare the effectiveness of using an onsite behavioral health specialist for screening, intervention and referral with basic written information and staff recommendations typically provided in primary care offices.

DETAILED DESCRIPTION:
There will be approximately 3-5 sites who will participate in this study. These sites may include two private practices in Roxboro and Creedmoor, North Carolina, the Duke Hospital and two practices in the Five County region of NC who are implementing Integrated, Collaborative, Accessible, Respectful, and Evidence-based (ICARE). In each clinic one day of the week (or 2 half days) will be chosen randomly from the days the clinic identifies as appropriate. During this time a behavioral health specialist (BHS) will be on site to recruit potential participants. All patients will be asked to speak to the specialist. On two other randomly selected days printed material will be given to all parents of underage patients and the underage patients. This material will describe the study and give the specialist's contact information. If the patients are 18 to 21 years old the material will be given directly to the patient.

The BHS will ask all interested participants to sign the informed consent/minor consent and one parent/legal guardian will be asked to counter sign the informed consent if subject is not 18 years of age yet. All participants signing informed consent will be given the CRAFFT and the PARTNER basic information questions in an interview with the specialist.

The primary outcome measure will be the number of participants recruited per day by the on site BHS versus appointment recruitment method. In addition, the total number of clinic visits for patients' ages 14 to 21 years old on each day of the week will be totaled by age, gender and ethnicity to determine the penetration rates for the recruitment procedures. And lastly, medical records at the treatment referral sites will be checked to identify the number of participants referred.

The study will recruit subjects at each site for approximately last six months.

ELIGIBILITY:
Inclusion Criteria:

Ages 12 through 20.

Exclusion Criteria:

None

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-02 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The trial will compare the effectiveness of using an onsite behavioral health specialist for screening, intervention and referral with basic written information and staff recommendations typically provided in primary care offices. | Same day

SECONDARY OUTCOMES:
Assessments and early intervention of identifying alcohol abuse in minors. | Same day

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Hubbard, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States